CLINICAL TRIAL: NCT00131157
Title: A Randomized-Controlled Evaluation of Spirometry Expert Support in General Practice
Brief Title: Evaluation of Spirometry Expert Support in General Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Boehringer Ingelheim (Industry); The Netherlands Asthma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 95500; NAF-3.4.02.18; ZonMW 920-03-265
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma; Cough; Dyspnea
Keywords: Pulmonary Disease, Chronic Obstructive; Family Practice; Spirometry; Decision Support Systems; Feedback
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Cough; Dyspnea

INTERVENTIONS:
Procedure: expert support for interpretation of spirometry

SUMMARY:
More and more general practitioners (GPs) use spirometry in their practices. At this time, there is sufficient reason to presume that, after a single postgraduate training program without any further support, most GPs have insufficient knowledge and ability to assure valid interpretation of their spirometry tests. Therefore, some kind of continuous diagnostic support with regard to spirometry interpretation by GPs is advisable. The aim of the present study is to assess whether implementation of spirometry expert support (either by a computerised expert system or a working agreement between general practitioners and respiratory consultants with respect to spirometry interpretation) causes changes in diagnosing and appropriateness and efficiency of medical care in subjects with chronic respiratory morbidity managed in general practice.

DETAILED DESCRIPTION:
More and more general practitioners (GPs) use spirometry in their practices. At this time, there is sufficient reason to presume that, after a single postgraduate training program without any further support, most GPs have insufficient knowledge and ability to assure valid interpretation of their spirometry tests. Therefore, some kind of continuous diagnostic support with regard to spirometry interpretation by GPs is advisable. The problem formulation for the study proposed is: "Does implementation of spirometry expert support (either by a computerized expert system or a local working agreement between GPs and respiratory consultants with respect to spirometry interpretation) cause changes in diagnosing and quality and efficiency of medical care in subjects with chronic respiratory morbidity managed in general practice?". In order to address this issue, two separate studies with different designs are proposed. Study I (n=62 GPs) is an 'in-depth' study of the GPs' decision-making process with regard to spirometry, and the impact of a computerized expert system on this process. Study II (n=39 general practices) is a pragmatic randomised-controlled implementation study evaluating two realistic modes of spirometry expert support (i.e., a computerized expert system or a working agreement between GPs and respiratory consultants).

ELIGIBILITY:
Inclusion Criteria:

* GP practices with a Windows supported electronic Patient Journal System (PJS) in a certain postal region in the Netherlands.

Exclusion Criteria:

* GP practices without a Windows supported PJS
* Practices outside a certain postcode region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2003-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Study I: between-group difference in the proportion of cases in which the GP opts for the gold standard diagnosis before versus expert/sham information
Study II: between-group difference in the proportion of patients with a changed respiratory diagnosis after spirometry interpretation in a random sample (n=20 patients) taken from an index population per practice

SECONDARY OUTCOMES:
Study I: between-group difference in the proportion of cases in which the GP opts for the gold standard treatment (prescription, referrals) before versus after the addition of expert/sham information
Study II: between-group difference in the proportion of ordered additional investigations and referrals by GPs

CONTACTS AND LOCATIONS:
Overall Officials: Chris van Weel, Prof, Principal Investigator — Radboud University Nijmegen Medical Centre, Nijmegen
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Chavannes N, Schermer T, Akkermans R, Jacobs JE, van de Graaf G, Bollen R, van Schayck O, Bottema B. Impact of spirometry on GPs' diagnostic differentiation and decision-making. Respir Med. 2004 Nov;98(11):1124-30. doi: 10.1016/j.rmed.2004.04.004. PMID 15526814
- [Background] Schermer TR, Jacobs JE, Chavannes NH, Hartman J, Folgering HT, Bottema BJ, van Weel C. Validity of spirometric testing in a general practice population of patients with chronic obstructive pulmonary disease (COPD). Thorax. 2003 Oct;58(10):861-6. doi: 10.1136/thorax.58.10.861. PMID 14514938
- [Derived] Poels PJ, Schermer TR, Thoonen BP, Jacobs JE, Akkermans RP, de Vries Robbe PF, Quanjer PH, Bottema BJ, van Weel C. Spirometry expert support in family practice: a cluster-randomised trial. Prim Care Respir J. 2009 Sep;18(3):189-97. doi: 10.4104/pcrj.2009.00047. PMID 19649513